CLINICAL TRIAL: NCT06238466
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD1705 Following Single and Multiple Ascending Doses in Participants With Dyslipidemia
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD1705 in Participants With Dyslipidemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D7650C00001
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular
Keywords: Dyslipidemia; Pharmacokinetics
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A1 (AZD1705) (Active Comparator): Non-Asian participants will receive AZD1705 subcutaneously on Day 1.
  Interventions: Drug: AZD1705
- Part A2 (AZD1705) (Active Comparator): Japanese participants will receive AZD1705 subcutaneously on Day 1.
  Interventions: Drug: AZD1705
- Part A3 (AZD1705) (Active Comparator): Chinese participants will receive AZD1705 subcutaneously on Day 1.
  Interventions: Drug: AZD1705
- Part B1 (AZD1705) (Active Comparator): Non-Asian participants who may or may not be receiving moderate- or high-intensity statin therapy will receive AZD1705 subcutaneously on Day 1 and Day 29.
  Interventions: Drug: AZD1705
- Part B2 (AZD1705) (Active Comparator): Japanese participants not receiving statin therapy will receive AZD1705 subcutaneously on Day 1 and Day 29.
  Interventions: Drug: AZD1705
- Part B3 (AZD1705) (Active Comparator): Participants who may or may not be receiving moderate- or high-intensity statin therapy and with the additional diagnosis of type 2 diabetes will receive AZD1705 subcutaneously on Day 1 and Day 29.
  Interventions: Drug: AZD1705
- Part A1 (Placebo) (Placebo Comparator): Non-Asian participants will receive placebo on Day 1.
  Interventions: Other: Placebo
- Part A2 (Placebo) (Placebo Comparator): Japanese participants will receive placebo on Day 1.
  Interventions: Other: Placebo
- Part A3 (Placebo) (Placebo Comparator): Chinese participants will receive placebo on Day 1.
  Interventions: Other: Placebo
- Part B1 (Placebo) (Placebo Comparator): Non-Asian participants who may or may not be receiving moderate- or high-intensity statin therapy will receive placebo on Day 1 and Day 29.
  Interventions: Other: Placebo
- Part B2 (Placebo) (Placebo Comparator): Japanese participants not receiving statin therapy will receive placebo on Day 1 and Day 29.
  Interventions: Other: Placebo
- Part B3 (Placebo) (Placebo Comparator): Participants who may or may not be receiving moderate- or high-intensity statin therapy and with the additional diagnosis of type 2 diabetes will receive placebo on Day 1 and Day 29.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD1705 — Participants will receive AZD1705 subcutaneously on Day 1 in Part A, and Days 1 and 29 in Part B.
  Arms: Part A1 (AZD1705); Part A2 (AZD1705); Part A3 (AZD1705); Part B1 (AZD1705); Part B2 (AZD1705); Part B3 (AZD1705)
Other: Placebo — Participants will receive placebo on Day 1 in Part A, and Days 1 and 29 in Part B.
  Arms: Part A1 (Placebo); Part A2 (Placebo); Part A3 (Placebo); Part B1 (Placebo); Part B2 (Placebo); Part B3 (Placebo)

SUMMARY:
A study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of AZD1705 in participants with dyslipidemia.

DETAILED DESCRIPTION:
This is a first time in human study in male and female (of non-childbearing potential) participants with dyslipidemia. The study consists of two parts:

1. Part A (single ascending dose): Part A of the study will include three parts: A1 for non-Asian participants, A2 for Japanese participants, and A3 for Chinese participants. Parts A2 and A3 are optional.
2. Part B (multiple ascending dose): Part B of the study will include three parts: B1 for non-Asian participants who may or may not be receiving moderate- or high-intensity statin therapy, B2 for Japanese participants not receiving statin therapy, and B3 for participants who may or may not be receiving moderate- or high-intensity statin therapy, with the additional diagnosis of type 2 diabetes (T2D), and with HbA1c < 8%. Parts B2 and B3 are optional.

The study will comprise of:

* A Screening Period of maximum 60 days for both Part A and Part B.
* Part A: A single dose of AZD1705 with an in-clinic period of 3 days.
* An outpatient Follow-up Period of approximately 16 weeks.
* Part B: 2 doses of AZD1705, given 28 days apart with an in-clinic period.
* An outpatient Follow-up Period of approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of non-childbearing potential participants with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test.
* Participants with elevated lipids.
* BMI between 18 and 35 kg/m^2.

Part B1 - May or may not be receiving moderate- or high-intensity statin therapy.

Part B3

* May or may not be receiving moderate- or high-intensity statin therapy.
* Diagnosed with T2D with hemoglobin A1c (HbA1c) < 8% level.

Parts B1 and B3

- Participants on medications should be on stable medication for ≥ 3 months before Screening with no planned medication or dose change during study participation.

Parts A2 and B2:

- Participants are to be Japanese, defined as having both parents and 4 grandparents who are Japanese.

Part A3:

- Participants are to be Chinese, defined as having both parents and 4 grandparents who are Chinese.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any laboratory values with the following deviations at the Screening Visit or on admission to the Clinical Unit. Abnormal values may be repeated once at the discretion of the Investigator:

  1. Alanine aminotransferase > 1.5 × upper limit of normal (ULN).
  2. Aspartate aminotransferase > 1.5 × ULN.
  3. Total bilirubin > ULN (Gilbert's syndrome).
  4. Estimated glomerular filtration rate < 60 milliliter (mL)/minute/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation 2021 (National Kidney Foundation).
  5. Hemoglobin < lower limit normal (LLN).
* Any clinically important abnormalities in hematology, coagulation, clinical chemistry, or urinalysis results other than those described under exclusion criterion number 4, at Screening and/or first admission to the study unit, as judged by the Investigator. Abnormal values may be repeated once at the discretion of the Investigator.
* Any positive result at Screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis C virus antibody (HCV Ab), or Human immunodeficiency virus (HIV).
* Abnormal vital signs, after 5 minutes supine rest, at Screening and/or first admission to the study unit, defined as any of the following:

  1. Systolic blood pressure (BP) ≤ 90 millimeters of mercury (mmHg) or > 140 mmHg (Part A) or > 150 mmHg (Part B).
  2. Diastolic BP < 50 mmHg or > 90 mmHg.
  3. Heart rate < 45 or > 90 beats per minute (bpm). Note: Blood pressure will be measured in triplicates and the mean value will be used. Where the values are outside the required range at admission, then based on medical history, one retest may be performed at this visit.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead ECG, at Screening and/or first admission to the study unit, as judged by the Investigator, that may interfere with the interpretation of QT interval corrected for heart rate (QTc) interval changes, including abnormal ST-T-wave morphology, particularly in the protocol-defined primary lead or left ventricular hypertrophy.

  1. Prolonged ECG interval measured from the onset of the QRS complex to the end of the T wave (QT) corrected for heart rate using Fridericia's correction (QTcF) > 450 ms.
  2. Family history of long QT syndrome.
  3. Time from the onset of the P wave to the start of the QRS complex (PR) (PQ) interval shortening < 120 milliseconds (ms) (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
  4. PR (PQ) interval prolongation (> 220 ms), persistent or intermittent second-degree atrioventricular (AV) block (participants with Wenckebach block while asleep are acceptable), third-degree AV block, or AV dissociation.
  5. Persistent or intermittent complete Bundle branch block (BBB), Intermittent bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with ECG interval measured from the onset of the QRS complex to the J point (QRS) > 110 ms.
* Participants with QRS > 110 ms but < 115 ms (Part A) or < 120 ms (Part B) are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
* Smokers who smoke > 10 cigarettes/day and are unable to comply with the nicotine restriction during the study.
* Known or suspected history of alcohol or drug abuse or those who consume > 3 units of alcohol per day for males or > 2 units of alcohol per day for females (where 1 unit being equal to approximately half pint [284 mL] of beer, one small glass [125 mL] of wine, or one measure [25 mL] of spirits) as judged by the Investigator.
* Positive screen for drugs of abuse or alcohol at Screening or on each admission to the Clinical Unit.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to study compound.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) defined as the regular consumption of more than 500 mg of caffeine per day (one cup ~100 mg caffeine; one cup of tea ~30 mg caffeine) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of investigational medicinal product (IMP). The period of exclusion begins after the final dose.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the Clinical Unit).
* Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Participants who are vegans or have medical dietary restrictions.
* Participants who cannot communicate reliably with the Investigator.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening or on admission as per site standard practice.
* Low-density lipoprotein (LDL) or plasma apheresis within 12 months prior to randomization.

Part A Only:

* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose), and minerals during the 2 weeks prior to the first administration of study intervention or longer if the medication has a long half-life.
* On statin therapy.
* Urine albumin: creatinine ratio > 30 mg/g.

Part B Only:

* Use of any herbal remedies, mega dose vitamins, and minerals during the two weeks prior to the first administration of study intervention or 5 half-lives, whichever is longer.
* Urine albumin: creatinine ratio > 100 mg/g.

Parts B1 and B3 Only:

- Contraindication to Magnetic Resonance Imaging (MRI) such as: participants with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field; participants with a history of extreme claustrophobia; or participants who cannot fit inside the MRI scanner cavity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Part A: From Screening (Day -60 to Day -2) until Day 113. Part B: From Screening until Day 141
  To assess the safety and tolerability of AZD1705 following subcutaneous administration of single ascending doses (Part A) and multiple ascending doses (Part B) in participants with dyslipidemia

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from zero extrapolated to infinity (AUCinf) | Part A: Day 1 to 113. Part B: Day 1 to 141
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Part A: Day 1 to 113. Part B: Day 1 to 141
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Maximum observed plasma (peak) drug concentration (Cmax) | Part A: Day 1 to 113. Part B: Day 1 to 141
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Cumulative amount of drug excreted unchanged (Ae) | Part A: Day 1 to 4. Part B: Day 1 to 4, and 29 to 30
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Fraction of drug excreted unchanged (fe) | Part A: Day 1 to 4. Part B: Day 1 to 4, and 29 to 30
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Rate of renal clearance of drug (CLR) | Part A: Day 1 to 4. Part B: Day 1 to 4, and 29 to 30
  To characterize the single and repeated dose PK of AZD1705 following subcutaneous administration in participants with dyslipidemia.
Change from baseline in target plasma protein | Part A: Baseline to Day 113. Part B: Baseline to Day 141
  To assess the effect of single and repeated subcutaneous AZD1705 administration on target plasma protein levels in participants with dyslipidemia.
Change from baseline in low-density lipoprotein cholesterol (LDL-C) | Part A: Baseline to Day 113. Part B: Baseline to Day 141
  To assess the effect of single and repeated subcutaneous AZD1704 administration on levels of LDL-C in circulation in participants with dyslipidemia.
Change from baseline in Apolipoprotein B (ApoB) | Part A: Baseline to Day 113. Part B: Baseline to Day 141
  To assess the effect of single and repeated subcutaneous AZD1704 administration on levels of ApoB in circulation in participants with dyslipidemia.
Change from baseline in triglycerides | Part A: Baseline to Day 113. Part B: Baseline to Day 141
  To assess the effect of single and repeated subcutaneous AZD1704 administration on levels of triglycerides in circulation in participants with dyslipidemia.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Glendale, California
  - Research Site, Jacksonville, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/